CLINICAL TRIAL: NCT05226611
Title: The Effect of Counterstrain Technique on Muscle Stiffness and Pain on Trapezius Tender Points in Medical Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #BHS-1561
Record Dates: First submitted 2022-01-12; First posted 2022-02-07 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Counterstrain; MyotonPRO; Tender Points
Keywords: Counterstrain; MyotonPRO; Tender points; Medical Students

STUDY DESIGN:
Masking Description: The participant felt which side was being treated however, the investigator measuring the physiologic parameters of the muscle with the MyotonPRO was blinded in terms of what side was being treated.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tender point treatment with Counterstrain (Experimental): A tender point was located in the upper trapezius region of the test subject and treated with counterstrain. The side with the highest initial pain level was used as the treatment side. Pain level was measured before and after treatment. The MyotonPRO was also used to measure physiologic parameters of the muscle before and after treatment.
  Interventions: Other: Counterstrain

INTERVENTIONS:
Other: Counterstrain — Counterstrain is a hands-on OMM technique that involves shortening the muscle to resolve the dysfunctional muscle stretch reflex and holding it for 90 seconds. The patient is then brought back to a neutral position and reassessed.

SUMMARY:
Medical students are prone to developing neck pain due to prolonged studying and poor posture. This can manifest as tender points in the upper trapezius region. Counterstrain (CS) is an osteopathic manipulative technique that has shown efficacy in previous studies in treating tender points. The MyotonPRO is a myotonometric device that can be used to measure various muscle parameters such as muscle stiffness. There is limited research regarding the use of osteopathic manipulative medicine to produce measurable changes in muscle stiffness by the MyotonPRO. This educational study aims to establish the efficacy of CS technique in decreasing the pain level of upper trapezius tender points in medical students as well as determining if CS causes a significant decrease in muscle stiffness in treated tender points as measured by the MyotonPRO. The investigators hope this educational study will encourage further studies on how osteopathic manipulative techniques affects the physiologic parameters of muscles.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age

Exclusion Criteria:

* Traumatized (sprained or strained) tissues, which would be negatively affected by the positioning of the patient
* Illness or other conditions in which strict positional restrictions preclude treatment
* Instability of the area being positioned that has the potential to produce unwanted neurologic or vascular side effects
* Vascular or neurologic syndromes, such as basilar insufficiency or neural foraminal compromise whereby the position of treatment has the potential to exacerbate the condition
* Severe degenerative spondylosis with local fusion and no motion at the level where treatment positioning would normally take place
* Pregnancy
* Positive for COVID-19 as well as symptoms indicating a SARS-CoV-2 infection

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-04-14 (Actual); Study Completion 2021-04-14 (Actual)

PRIMARY OUTCOMES:
Pain level | This was done immediately before and immediately after counterstrain treatment. Counterstrain treatment is a hands-on osteopathic manipulative technique that involves shortening the muscle belly of the painful region.
  Pain level of the tender point as rated by the test subject out of a scale of 1 to 10, 1 being very little pain and 10 being the most pain the test subject has ever felt.

SECONDARY OUTCOMES:
Muscle Stiffness | This was done immediately before and immediately after counterstrain treatment. Counterstrain treatment is a hands-on osteopathic manipulative technique that involves shortening the muscle belly of the painful region.
  Muscle stiffness measured by the MyotonPRO, a myotonometric device that applies a brief mechanical impulse to the targeted muscle, used to measure physiologic parameters such as muscle stiffness.

CONTACTS AND LOCATIONS:
Locations (1):
- NYIT College of Osteopathic Medicine, Glen Head, New York, United States

IPD SHARING:
Plan to Share IPD: No